CLINICAL TRIAL: NCT01450085
Title: Impact of a New Molecular Tuberculosis (TB) Test on TB/HIV Outcomes Among HIV-
Brief Title: Chepetsa TB - Reducing TB Among HIV-Infected Malawians
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1R01AI093316-01A1 (NIH)
Record Dates: First submitted 2011-10-07; First posted 2011-10-12 (Estimated); Last update posted 2017-08-18 (Actual); Status verified 2017-08

CONDITIONS: Tuberculosis
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GeneXpert (Active Comparator): Point of care GeneXpert
  Interventions: Other: GeneXpert; Other: LED Microscopy
- LED Microscopy (Active Comparator): Point of care LED Microscopy
  Interventions: Other: LED Microscopy

INTERVENTIONS:
Other: GeneXpert — Point of care GeneXpert
  Arms: GeneXpert
Other: LED Microscopy — Point of care LED Microscopy

SUMMARY:
The specific aims of this project are: (1) to compare the impact of using the routine screening and GeneXpert algorithms for TB case detection on Tuberculosis (TB)- and HIV-related outcomes; (2) to compare the impact of using the routine screening and GeneXpert algorithms for exclusion of TB prior to initiation of IPT and ART on TB- and HIV-related outcomes; and (3) to assess the relative cost-effectiveness of the routine screening and GeneXpert algorithms for TB case detection and exclusion of TB. The GeneXpert is a "disruptive technology"10 that could allow TB/HIV programs in resource-limited settings to leapfrog over solid and liquid culture-based TB diagnostic algorithms, and to remove a key barrier to scale up of ICF and IPT.

DETAILED DESCRIPTION:
HIV and tuberculosis (TB) are, along with malaria, the leading infectious causes of death worldwide and in sub-Saharan Africa.1 In 2008, there were 2 million deaths from AIDS and 1.8 million deaths from TB worldwide.2, 3 The HIV epidemic has fueled an increase in the incidence of, prevalence of and mortality due to TB in the past 3 decades. 15% of TB cases are HIV co-infected worldwide.34 78% of HIV-infected TB cases are in Africa.3 TB is the leading cause of death and opportunistic infection among persons living with HIV/AIDS (PLWHA). The HIV epidemic has challenged time-tested TB control methods that are now failing in high HIV prevalence settings.5 The World Health Organization (WHO) has recommended that the Three I's - intensified case-finding for TB (ICF), isoniazid preventive therapy (IPT) and infection control for TB - be targeted at PLWHA.6 ICF and IPT have not been adequately implemented in part due to the absence of sensitive, specific and rapid TB tests. The Cepheid GeneXpert System, a new diagnostic test for TB, is a self-contained sputum-processing and real-time PCR system to detect the M. tuberculosis complex as well as rifampin resistance.78 The GeneXpert is rapid, highly sensitive and specific, can be used as a point-of-care test, and has low human resource, laboratory and infection control requirements.7, 8 The WHO Strategic and Advisory Group for TB has endorsed recommendations for widespread use of the GeneXpert.9 WHO strongly recommended that the GeneXpert should be used as the initial diagnostic test in HIV-infected TB suspects and multidrug-resistant TB (MDR-TB) suspects.9 WHO also recommended that implementation of the GeneXpert be phased in within the context of comprehensive national and MDR-TB strategic plans.9 WHO recognized that several operational conditions need to be met for successful implementation, including but not limited to stable electrical supply, security against theft, trained personnel and annual calibration of the instrument by a commercial supplier.9 WHO also noted that it is important to document the impact and cost-effectiveness of the GeneXpert for TB case detection.9

Trial Concept The overall objective of this proposal is to conduct a cluster-randomized trial of the relative impact and cost-effectiveness of a routine TB screening algorithm -- symptom screening and point-of-care LED fluorescence sputum smear microscopy - versus a GeneXpert-based TB screening algorithm - symptom screening and point-of-care GeneXpert testing - on reducing morbidity and mortality due to TB among HIV-infected Malawians. 12 public sector clinics in southern Malawi will be randomized to 1 of 2 algorithms for TB case detection as part of ICF and for exclusion of TB prior to IPT and antiretroviral therapy (ART) initiation. In the clinics assigned to the GeneXpert algorithm, newly diagnosed HIV-infected patients will be screened for symptoms of TB and, if symptomatic, will provide sputum for GeneXpert point-of-care TB testing. Under the routine screening algorithm, patients at a clinic will be screened for symptoms of TB and, if symptomatic, will provide sputum for point-of-care LED fluorescence smear microscopy. The current standard of care in Malawi and most of Africa is symptom screening and sputum smear microscopy using Ziehl-Neelsen stain (not LED fluorescence microscopy) alone. There is not sufficient evidence at this time to demonstrate whether point-of-care LED microscopy versus GeneXpert testing is likely to be superior with respect to clinical impact and/or cost-effectiveness. Outcomes will be measured at the clinic level.

ELIGIBILITY:
Inclusion Criteria:

All HIV-infected men and women > 18 years of age with newly diagnosed HIV at the 12 study clinics will be asked to participate in the study.

Exclusion Criteria:

* Patients will be excluded from participation if they have a current diagnosis of TB and/or if they are currently taking IPT, TB treatment and/or ART.
* Patients will also be excluded from participation if they cannot speak English or Chichewa;
* if they have a language or hearing impairment; or
* if they are prisoners.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Actual)
Dates: Start 2012-09; Primary Completion 2016-12 (Actual); Study Completion 2016-12-30 (Actual)

PRIMARY OUTCOMES:
Survival of newly-diagnosed HIV-infected patients at 1 year | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Corbett, MD, Principal Investigator — Malawi Liverpool Wellcome Trust; David Dowdy, MD. PhD, Study Director — Johns Hopkins Unviversity; Lawrence Moulton, PhD, Principal Investigator — Johns Hopkins University
Locations (2):
- Malawi (2):
  - Blantyre, Thyolo District
  - Blantyre

REFERENCES:
- [Derived] Ngwira LG, Corbett EL, Khundi M, Barnes GL, Nkhoma A, Murowa M, Cohn S, Moulton LH, Chaisson RE, Dowdy DW. Screening for Tuberculosis With Xpert MTB/RIF Assay Versus Fluorescent Microscopy Among Adults Newly Diagnosed With Human Immunodeficiency Virus in Rural Malawi: A Cluster Randomized Trial (Chepetsa). Clin Infect Dis. 2019 Mar 19;68(7):1176-1183. doi: 10.1093/cid/ciy590. PMID 30059995
- [Derived] Ngwira LG, Dowdy DW, Khundi M, Barnes GL, Nkhoma A, Choko AT, Murowa M, Chaisson RE, Corbett EL, Fielding K. Delay in seeking care for tuberculosis symptoms among adults newly diagnosed with HIV in rural Malawi. Int J Tuberc Lung Dis. 2018 Mar 1;22(3):280-286. doi: 10.5588/ijtld.17.0539. PMID 29471905